CLINICAL TRIAL: NCT00416338
Title: Comparison of Two Exit-Site Care Methods, Film Dressing (F) Method and Simple Gauze Dressing (G) Method, in Chronic Peritoneal Dialysis (CPD) Patients
Brief Title: Method of Exit Site Care in Chronic Peritoneal Dialysis Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We encounter technical problems to continue with the study. (Notably difficulty in teaching the patients to use the dressing set involved in the study.)
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2006.401-T
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-04

CONDITIONS: Chronic Peritoneal Dialysis
Keywords: renal failure; infection; peritonitis
MeSH Terms: conditions — Renal Insufficiency; Infections; Peritonitis

INTERVENTIONS:
Device: film dressing by adhesive

SUMMARY:
Peritoneal dialysis accounts for more than 70% of the dialysis modality in Hong Kong. Exit site infection (ESI) is one of the causes leading to peritoneal catheter removal. Appropriate exit-site care can prevent ESI. As the presence of a causative organism is essential in ESI, eliminating organism invasion may be useful in preventing ESI. In the present study, an exit site care method aiming at preventing organism invasion is developed to investigate its effectiveness in reducing ESI. It is also hoped the present study can help to develop an exit site care method that can reduce the frequency of exit site dressing so as to reduce the burden of patients and to improve their quality of life.

We'll recruit one hundred new chronic peritoneal dialysis patients into the study. The patients will be divided into two groups. One group of the patients will use film-dressing method (F) and the other group will use simple gauze dressing method (G). F group patients will have the exit site covered with a dressing film and keep it intact for 7 days after having the exit site cleaned with antiseptic solution. G group patients will clean the exit site with antiseptic solution and change the simple gauze dressing daily.

The outcomes of the two groups will be compared. The outcome will be expressed in terms of exit site infection free period, peritonitis free period and exit site condition classification. Patient subjective quality of life will also be compared at first and twelfth month.

ELIGIBILITY:
Inclusion Criteria:

* chronic renal failure patients with peritoneal catheter newly inserted

Exclusion Criteria:

* Patients have exit-site infection before stitches removal or presence of signs and symptoms of exit-site infection at the time of remove stitches.
* Patients plan to move out of PWH or transplant soon after catheter insertion.
* Patients have known history of allergy to adhesives / tapes.
* Extremely non-compliant patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-01; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Exit site infection.

SECONDARY OUTCOMES:
Patient satisfaction / quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Man-Ching Law, BN, Principal Investigator — Renal Unit, Department of Medicine & Therapeutics, Prince of Wales Hospital, Hong Kong
Locations (1):
- Department of Medicine & Therapeutics, Prince of Wales Hospital, Shatin, Hong Kong